CLINICAL TRIAL: NCT02973347
Title: Impact of Intermittent and Continuous Enteral Feeding on Ventilator-associated Pneumonia in Pediatric ICUs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Children's Hospital of Fudan University (Other); Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XH-16-039
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Enteral Feeding; Ventilator-Associated Pneumonia
Keywords: Enteral Feeding; Ventilator-Associated Pneumonia; Mechanical Ventilation; Pediatric Intensive Care Unit; Critical Illness
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent enteral feeding (Active Comparator): Intermittent enteral feeding via the nasogastric tube is applied less than 30 mins.
  Interventions: Other: Intermittent enteral feeding
- Continuous enteral feeding (Active Comparator): Continuous enteral feeding via the nasogastric tube using infusion pump is applied for 24 hours.
  Interventions: Other: Continuous enteral feeding

INTERVENTIONS:
Other: Intermittent enteral feeding — The intervention is the schedule under which ventilated children are offered enteral feeding attempts: feed administered via the nasogastric tube less than 30 mins.
  Arms: Intermittent enteral feeding
Other: Continuous enteral feeding — The intervention is the schedule under which ventilated children are offered enteral feeding attempts: feed administered via the nasogastric tube for 24 hours.
  Arms: Continuous enteral feeding

SUMMARY:
Mechanical ventilation has become one of the most important supportive treatment methods to save the life of critically ill children over time. Ventilator-associated pneumonia (VAP) is a common complication of mechanical ventilation. It is one of the leading causes of hospital-acquired infections in the Paediatric Intensive Care Unit (PICU).VAP can aggravate patients' condition and have adverse effect on mechanical ventilation. Moreover, VAP is associated with significant increased mortality. In those critical ill patients, the catabolism increased, the anabolism decreased, which can induce negative nitrogen balance. The consensus of optimal nutrition therapy in pediatric critical care in the Asia-Pacific, released in 2014, clearly recommended that early enteral nutrition support, which begin within 24-48 hours after admitting in PICU, can significantly reduce the prevalence and mortality of nosocomial infection. Intermittent enteral feeding and continual enteral feeding are the most common methods of enteral nutrition at present. There is no final conclusion about the association between enteral nutrition methods and VAP. Thus, the relationship between enteral feeding and VAP has long been a controversial issue. There is little clinical research on the correlation between enteral nutrition and VAP in children with mechanical ventilation, and mostly were observational studies which lacks strong evidence. How to choose the appropriate enteral nutrition remains an urgent need in PICU clinical work. Therefore, it is necessary for us to analyze the relationship between enteral feeding and VAP in critically ill children. This study would perform a two-year research with mechanical ventilated patients in PICU of four children hospitals in Shanghai, which aim to determine the relationship between different enteral feeding methods and VAP, to collect the baseline characteristic data of ventilated children, to analyze the risk factors for VAP in PICU patients. The results from our study would contribute to improving the standard of care for children undergoing mechanical ventilation, reducing their lung injury and improving prognosis.

DETAILED DESCRIPTION:
With the development and advancement of modern medical technology, mechanical ventilation has become one of the most important supportive treatment methods to save the life of critically ill children. Ventilator-associated pneumonia （VAP） is a common complication of mechanical ventilation. It is one of the leading causes of hospital-acquired infections in the PICU. VAP can aggravate patients' condition and have adverse effect on mechanical ventilation. An overseas study reported that VAP increased 56% of the PICU length of stay and 43% of the length of hospitalization. Moreover, VAP is associated with significant increased mortality. Because the prevalence and mortality of VAP vary in adult and children, also in different area, it is very necessary to investigate the current status of VAP in local children, which can contribute to clinical prevention and treatment to decrease mortality. Appropriate nutrition support can improve the body's metabolism, promote tissue and body function repair, reduce the incidence of complications. However, inadequate enteral nutrition may cause gastroesophageal reflux and aspiration, which may lead to VAP and exacerbate the condition. Intermittent enteral feeding and continual enteral feeding are the most common methods of enteral nutrition at present. The relationship between enteral feeding methods and VAP has long been a controversial issue. There is little clinical research on the correlation between enteral feeding and VAP in children with mechanical ventilation, and mostly were observational studies which lacks strong evidence. How to choose the appropriate enteral nutrition remains an urgent need in PICU clinical work. Therefore, it is necessary for us to analyze the relationship between enteral feeding and VAP in critically ill children.

The primary objective of this study is to investigate the influence of intermittent or continuous enteral feeding on VAP in PICUs. The secondary objectives are to collect the baseline characteristic data of ventilated children, and to analyze the risk factors of VAP in children. Each patient will be randomly assigned to an intermittent or continuous enteral feeding schedule. Intermittent enteral feeding schedule: feed administered via the nasogastric tube less than 30 mins. Continuous enteral feeding schedule: feed pump delivered via the nasogastric tube over 24 hours. Data on feeding progression, respiratory status and incidence of VAP will be collected and compared. The study will also collect data on baseline characters, ventilation management, ventilated days and the time to discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age of 29 days to 16 years.
* Subjects ventilated over or equal to 12 hours.
* Endotracheal intubation.
* Subjects without contraindication for enteral feeding.

Exclusion Criteria:

* Newborn or age > or equal to 16 years.
* Subjects has been ventilated before this research.
* Subjects ventilated less than 12 hours.
* Invasive ventilation.
* Subjects with severe congenital malformations.

Ages: 29 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Ventilator-associated pneumonia | at Day-28
  The incidence of VAP in patients with intermittent enteral feeding strategy is compared with the incidence of VAP in patients with continuous enteral feeding strategy. Diagnosis of VAP as defined by national diagnostic criteria.

SECONDARY OUTCOMES:
Duration of ICU stay | at Day-28
Duration of hospital stay | at Day-28
ICU mortality | at Day-28
Hospital mortality | at Day-28

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhu, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Yueniu Zhu, PhD, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided